CLINICAL TRIAL: NCT04976790
Title: Effectiveness, Safety and Economic Evaluation of Chinese Tuina (Chinese Massage and Flurbiprofen Cataplasms) in the Treatment of Chronic Nonspecific Low Back Pain
Brief Title: Chinese Tuina Therapy for Treatment of Chronic Nonspecific Low Back Pain
Acronym: CNLBPCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Changhe Yu, Clinical professor, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021DZMEC-070-01
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Chronic Nonspecific Low Back Pain
Keywords: Massage; Tuina; Traditional Chinese medicine; CEA; CUA; ICER

STUDY DESIGN:
Intervention Model Description: Two arms recruit and evaluate the participants at the same time, and the included participants have the equal opportunity to either the Chinese Tuina or the Flurbiprofen Cataplasms treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese Tuina group (CTG) (Experimental): The participants in Chinese Tuina group will receive the traditional Chinese Tuina therapy on the basis of health education and home-exercise. All the treatment will cost 20-25 minutes. Patients in this group received 4 treatments over 14 days.
  Interventions: Behavioral: Chinese Tuina therapy
- Flurbiprofen Cataplasms group (FCG) (Active Comparator): The FCG group received flurbiprofen gel on the basis of the health education and home-exercise, twice daily, for 14 days.
  Interventions: Drug: Flurbiprofen Cataplasms group (FCG).

INTERVENTIONS:
Behavioral: Chinese Tuina therapy — Firstly, the patient is in the prone position, and the doctor use the method of rolling or kneading the Bladder meridians on both sides of the spine. The waist will be focused on to manipulate preferentially and then using the same technique on the patient's back, buttocks and lower limbs. Secondly, the physician will perform the manipulation on the patient's waist and the posterolateral side of the lower limbs by pressing, kneading, plucking. The doctors press the acupoints, including Mingmen(DU04),Shenshu(BL23),Yaoyangguan(DU03),Huantiao(GB30), Weizhong(BL40),Chengshan(BL57),and Ashi points, with the elbow or the thumb to achieve Deqi sensation. Thirdly, the The doctor uses the method of pressing acupoints, including Tianshu(ST25),Qichong(ST30),Chongmen(SP12),Daimai(GB26),Jingmen(GB25) on both sides. Fourthly, the patient is required to face the doctor in a lateral position for pulling manipulation on the both sides of lumbar vertebrae.
  Arms: Chinese Tuina group (CTG)
Drug: Flurbiprofen Cataplasms group (FCG). — One Flurbiprofen Cataplasm was applied to the left and right sides of the waist, twice daily, for 14 days
  Other Names: ZePuSi
  Arms: Flurbiprofen Cataplasms group (FCG)

SUMMARY:
Chronic Nonspecific Low back Pain (NLBP) is a common symptom in today's society. It causes serious health and economic burdens. Low back pain can be attributed to excessive physical exertion or trauma, resulting in damage or degradation of the vertebrae, intervertebral discs, or spinal muscles and nonspecific low back pain typically can account for 90% of the patients with 35 to 55 years old. Some guidelines endorse the cautious use of medication and surgery and take nonpharmacological and noninvasive treatments as a first-line treatment, including routine health education, exercise, psychotherapy, and physical therapies, owing to the risk of trauma and the cost. With a long history, Tuina is a one of the common nonsurgical methods to treat LBP in China.. The effect of Tuina is attributed to relaxing muscles and tendons, improving circulation, regulating spinal balance, decreasing edema and aseptic inflammation. Many clinical reports have confirmed its effectiveness, but more clinical trials are required to provide evidence of Tuina for low back pain. Therefore, this study was designed to compare the effectiveness of Tuina with Flurbiprofen Cataplasms for patients with low back pain on the basis treatment of health education and self-management exercise at home.

DETAILED DESCRIPTION:
This study is a single-center, assessor- and analyst-blinded randomized controlled trial conducted in Beijing, China, at Dongzhimen hospital affiliated to Beijing university of Chinese medicine. In total, 90 patients will be recruited and randomly assigned to a Tuina group and a Flurbiprofen Cataplasms group in a 1:1 ratio. The Chinese Tuina group will be given twice per week for 14 days, and medicine group will be given Flurbiprofen Cataplasms twice daily for 14 days. We will ask some researchers who are blinded to assignment to accomplish the outcome assignment and statistical analyses independently. The outcome will be measured by three self-report questionnaires, which can reflect the lumbar dysfunction, pain, quality of life, and adverse events. Four time points will be used to assess outcomes, including baseline, 7 days, 14 days and 28 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-specific low back pain;
* Aged between 18 and 65,male and female;
* Duration of low back pain as the main symptom for at least 12 weeks;
* pain intensity with NRS score equals or more than 4;
* X-ray or CT on low back helped to confirm no lumbar diseases;
* Ability to understand and complete the questionnaires;
* Any treatments aiming to CNLBP need more than 1 month washout period;
* Volunteer to participate in the study and informed consent form.

Exclusion Criteria:

* Sciatica, myelopathy, displacement, or radiculopathy due to lumbar intervertebral disc disorders or Spondylolisthesis；
* Chronic low back pain caused by local disease (e.g., lumbar fracture, lumbar tumor, lumbar tuberculosis, lumbar spine surgery or trauma)；
* Immune diseases such as rheumatoid joints and ankylosing spondylitis；
* Severe primary disease such as cardiovascular, lung, kidney, and hematopoietic disease;
* Pregnant or lactating women;
* patients with skin injury;
* Allergy or intolerance to Non-steroidal anti-inflammatory drug (e.g., asthma, gastrointestinal ulcers, and bleeding);
* Mental illness；
* Poor compliance of examination and treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Changes in NRS scores for pain intensity | Change from baseline at 14 days
  The changes in NRS scores at 14 days after randomization.

SECONDARY OUTCOMES:
Changes in NRS scores for pain intensity | Change from baseline at 7 days and 28 days after randomization
  The NRS scores are measured at baseline, 7 days and 28days after randomization
Changes in the ODI scores for lumbar function | Change from baseline at 7 days,14 days and 28 days after randomization
  The ODI (Oswestry Low Back Pain Disability Index) scores are measured at baseline, 7 days, 14 days and 28 days after randomization
Clinical effective rate | Change from baseline at 7days,14days and 28 days after randomization
  The clinical response rate is measured at baseline, 7 days, 14 days and 28 days after randomization
Changes in 7-level Likert Scale for patient assessment global improvement | Change from baseline at 7 days,14 days and 28 days after randomization
  The PAG with 7-level Likert Scale is measured at baseline, 7 days, 14 days and 28 days after randomization
Changes in PROMIS® Scale v1.2 Scale for patient assessment global improvement | Change from baseline at 14 days after randomization
  The PAG with PROMIS® Scale v1.2 Scale is measured at baseline, 14 days after randomization
Changes in the Quebec Low Back Pain Disability Scale scores for lumbar function | Change from baseline at 14 days after randomization
  The Quebec Low Back Pain Disability Scale scores are measured at baseline and 14 days after randomization
Changes in PROMIS® Item Bank v2.0-Physical Function scores for Physical Function | Change from baseline at 14 days after randomization
  The PROMIS® Item Bank v2.0-Physical Function-Short Form 8c 7-Day Scale scores are measured at baseline and 14 days after randomization
Changes in Quality adjusted life years (QALY) | Change from baseline at 7 days,14 days and 28 days after randomization
  The quality adjusted life years (QALY) of the subjects were measured by TCM health-related life quality scale (CM-QOL), five-dimensional health scale (EQ-5D) and SF-6D at baseline, 7 days, 14 days and 28 days after randomization
Incidence of adverse events | Change from baseline at 7 days,14 days and 28 days after randomization
  The incidence of adverse events during treatment will be calculated
Cost-Effectiveness Analysis (CEA) ratio | Change from baseline at 7 days,14 days and 28 days after randomization
  The cost-effectiveness ratio (C/E) is measured at baseline,7days,14 days and 28 days after randomization
Cost-utility analysis (CUA) ratio | Change from baseline at 7 days,14 days and 28 days after randomization
  The cost-utility ratio (C/U) is measured at baseline,7days,14 days and 28 days after randomization
Incremental cost-effectiveness ratio and Incremental cost-utility ratio | Change from baseline at 7 days,14 days and 28 days after randomization
  Incremental cost-effectiveness ratio and Incremental cost-utility ratio are measured at baseline,7days,14 days and 28 days after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Xiyou Wang, Principal Investigator — Beijing University of Chinese Medicine affiliated Dongzhimen Hospital
Locations (1):
- Beiing university of Chinese medicine Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No